CLINICAL TRIAL: NCT06875076
Title: Efficacy and Safety of Ivonescimab (AK112) in Combination with Chemotherapy for the Treatment of Pretreated Pleural Mesothelioma: a Phase II Multicenter, Single-Arm Clinical Trial
Brief Title: Multicenter Single-Arm Study of Ivonescimab (AK112) Combined with Chemotherapy in Pretreated Pleural Mesothelioma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Hospital of Jilin University (Other)
Responsible Party: Principal Investigator, Kewei Ma, Professor, The First Hospital of Jilin University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 24K353-001
Record Dates: First submitted 2025-03-08; First posted 2025-03-13 (Actual); Last update posted 2025-03-13 (Actual); Status verified 2025-03

CONDITIONS: Pretreated Pleural Mesothelioma
MeSH Terms: interventions — Drug Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- treatment (Experimental): ivonescimab 20mg/kg combined with pemetrexed 500mg/m²/gemcitabine 1000mg/m²/vinorelbine 25mg/m² every 21 days for 4 cycles followed by a maintenance phase (ivonescimab monotherapy 20mg/kg every 21 days until disease progression, intolerance, or up to 2 years).
  Interventions: Drug: Ivonescimab Combined With Chemotherapy

INTERVENTIONS:
Drug: Ivonescimab Combined With Chemotherapy — ivonescimab 20mg/kg combined with pemetrexed 500mg/m²/gemcitabine 1000mg/m²/vinorelbine 25mg/m² every 21 days for 4 cycles followed by a maintenance phase (ivonescimab monotherapy 20mg/kg every 21 days until disease progression, intolerance, or up to 2 years)

SUMMARY:
This study is a prospective, multicenter, single-arm, Phase II clinical trial evaluating the efficacy and safety of ivonescimab (AK112) combined with chemotherapy in patients with pleural mesothelioma who failed prior immunotherapy, anti-angiogenic therapy, or chemotherapy. The regimen consists of a treatment phase (ivonescimab 20mg/kg combined with pemetrexed 500mg/m²/gemcitabine 1000mg/m²/vinorelbine 25mg/m² every 21 days for 4 cycles) followed by a maintenance phase (ivonescimab monotherapy 20mg/kg every 21 days until disease progression, intolerance, or up to 2 years).The trial plans to enroll 25 patients, with the primary endpoint being objective response rate (ORR). Secondary endpoints include progression-free survival (PFS), overall survival (OS), and safety profiles. Exploratory endpoints investigate biomarkers such as tertiary lymphoid structures, tumor-infiltrating lymphocytes, and macrophage polarization within the tumor microenvironment.

DETAILED DESCRIPTION:
Study Protocol Overview This is a prospective, multicenter, single-arm Phase II clinical trial evaluating the efficacy and safety of ivonescimab (AK112) combined with chemotherapy in pretreated pleural mesothelioma patients who failed prior immunotherapy, anti-angiogenic therapy, or chemotherapy. Utilizing a Simon two-stage design, the study plans to enroll 25 participants. The primary endpoint is objective response rate (ORR), with secondary endpoints including progression-free survival (PFS), overall survival (OS), and safety profiles. Exploratory endpoints investigate biomarkers such as tertiary lymphoid structures, tumor-infiltrating lymphocytes, and macrophage polarization in the tumor microenvironment.

Treatment Regimen Treatment Phase: Ivonescimab (20mg/kg, Q3W) combined with chemotherapy (pemetrexed 500mg/m², gemcitabine 1000mg/m², or vinorelbine 25mg/m²) for 4 cycles.

Maintenance Phase: Ivonescimab monotherapy (20mg/kg, Q3W) until disease progression, intolerance, or up to 2 years.

Inclusion Criteria Asian ethnicity, aged 18-75, ECOG 0-1; Histologically confirmed malignant pleural mesothelioma; Progression after ≥1 and ≤2 prior systemic therapies (platinum-based chemotherapy, immunotherapy combinations, or anti-angiogenic therapy);

≥1 measurable lesion (modified RECIST 1.1); Adequate organ function (hemoglobin ≥90g/L, neutrophils ≥1.5×10⁹/L, creatinine clearance ≥50ml/min).

Exclusion Criteria History of other malignancies within 5 years (except cured skin carcinoma or in situ cancer); Tumor encasing critical vasculature or with necrosis/cavitation posing bleeding risks; Active hepatitis B (untreated HBV DNA≥1000 copies/ml), HIV, or HCV infection; Active autoimmune disease requiring systemic treatment within 2 years; Participation in other interventional studies within 4 weeks prior to enrollment.

Sample Size Calculation Based on Simon's two-stage design, assuming ORR improvement from 6% to 25% (α=0.05, power=80%). Stage 1 enrolls 9 patients; if ≤2 responses occur, the trial stops. Otherwise, Stage 2 proceeds, totaling 25 participants.

Study Endpoints Primary: Objective response rate (ORR); Secondary: PFS, OS, disease control rate (DCR), duration of response (DoR), safety; Exploratory: Tertiary lymphoid structures (CD3/CD20/CD21), tumor-infiltrating lymphocytes (CD4/FOXP3), macrophage polarization (M1:M2).

ELIGIBILITY:
Inclusion Criteria:

1. Asian ethnicity, aged 18-75, ECOG 0-1;
2. Histologically confirmed malignant pleural mesothelioma;
3. Progression after ≥1 and ≤2 prior systemic therapies (platinum-based chemotherapy, immunotherapy combinations, or anti-angiogenic therapy);
4. ≥1 measurable lesion (modified RECIST 1.1);
5. Adequate organ function (hemoglobin ≥90g/L, neutrophils ≥1.5×10⁹/L, creatinine clearance ≥50ml/min).

Exclusion Criteria:

1. History of other malignancies within 5 years prior to enrollment, except cured basal cell carcinoma, squamous cell carcinoma of the skin, or carcinoma in situ with radical resection. Patients diagnosed with other malignancies or lung cancer more than 5 years prior to enrollment require pathological/cytological confirmation of recurrent lesions.
2. Radiologically confirmed tumor encasement of major blood vessels, necrosis, or cavitation with significant bleeding risk as judged by the investigator.

   Tumor invasion of adjacent critical organs/vessels (e.g., heart/pericardium, trachea, esophagus, aorta, superior vena cava) or risk of esophageal-tracheal/pleural fistula.
3. Current participation in other interventional clinical trials or receipt of investigational drugs/devices within 4 weeks prior to the first dose.
4. Palliative local therapy for non-target lesions within 2 weeks prior to the first dose; non-specific immunomodulatory therapy (e.g., interleukin, interferon, thymosin, TNF-α, excluding IL-11 for thrombocytopenia) within 2 weeks; or herbal/Chinese patent medicines with anticancer indications within 1 week.
5. Prior systemic anti-angiogenic therapy combined with PD-1/PD-L1 inhibitors, including bevacizumab (and biosimilars), endostatin, small-molecule TKIs, ramucirumab, etc.
6. Bleeding history ≥ Grade 3 (CTCAE v5.0) within 4 weeks prior to screening. History of solid organ or hematopoietic stem cell transplantation.
7. Uncontrolled active infections (e.g., acute pneumonia) or acute exacerbation of chronic obstructive pulmonary disease within 1 month; active tuberculosis (TB) requiring clinical exclusion.
8. Idiopathic pulmonary fibrosis, organizing pneumonia (e.g., bronchiolitis obliterans), or drug-induced pneumonitis.
9. Major surgery or severe trauma within 30 days prior to the first dose, or planned major surgery within 30 days after the first dose; minor procedures (excluding PICC/port placement) within 3 days.
10. History of myocarditis, cardiomyopathy, or malignant arrhythmia; acute myocardial infarction, unstable angina, or NYHA Class III-IV heart failure within 12 months.
11. Uncontrolled hypertension (≥150/100 mmHg despite medication) or hypertensive crisis/encephalopathy.
12. Active central nervous system (CNS) metastases or carcinomatous meningitis, except asymptomatic brain metastases.
13. Active gastrointestinal bleeding, ulcers, or perforation risk (e.g., hematemesis ≥5 mL/day, melena, or hematochezia).
14. Active autoimmune diseases requiring systemic treatment (e.g., immunosuppressants/corticosteroids) within 2 years. Replacement therapies (e.g., thyroid hormone, insulin) are allowed.
15. Chronic corticosteroid use (>10 mg/day prednisone equivalent). Inhaled corticosteroids for asthma/COPD or topical steroids are permitted.
16. Non-healing wounds or unhealed fractures.
17. Known hypersensitivity to any study drug component or severe hypersensitivity to monoclonal antibodies.
18. Reproductive criteria:

    Female: Non-sterilized, non-menopausal, or unwilling to use contraception during and for 6 months post-treatment; positive pregnancy test or lactation.

    Male: Non-sterilized or unwilling to use contraception during and for 6 months post-treatment.
19. HIV infection (positive HIV1/2 antibodies).
20. Untreated active hepatitis B (HBV DNA ≥1000 copies/mL). Patients with HBV DNA <1000 copies/mL must receive antiviral therapy throughout the study.
21. Active HCV infection (positive HCV antibody with detectable HCV-RNA). Substance abuse or psychiatric disorders affecting compliance.
22. Live vaccination within 30 days prior to the first dose (inactivated vaccines allowed).
23. Other conditions that may interfere with study results, preclude full participation, or are deemed by the investigator to conflict with the subject's best interest.

Ages: 18 Months to 75 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 25 (Estimated)
Dates: Start 2025-03-08 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-12 (Estimated)

PRIMARY OUTCOMES:
objective response rate (ORR) | From enrollment to the end of treatment at 3 months

SECONDARY OUTCOMES:
progression-free survival (PFS) | From enrollment to the end of treatment at 3 years
overall survival (OS) | From enrollment to the end of treatment at 5 years
adverse effect | From enrollment to the end of treatment at 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Ma, Study Chair — The First Hospital of Jilin University
Locations (1):
- Cancer center, First Hospital of Jilin University, Changchun, Jilin, China